CLINICAL TRIAL: NCT03828799
Title: Safety, Tolerability and Efficacy of Regorafenib in Combination With FOLFIRINOX in Patients With RAS-mutated Metastatic Colorectal Cancer: a Dose-escalation, Phase I/II Trial
Brief Title: Safety, Tolerability and Efficacy of Regorafenib in Combination With FOLFIRINOX in Patients With Colorectal Cancer
Acronym: FOLFIRINOX-R
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2018-003541-42
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Colorectal cancer; Folfirinox; Regorafenib; RAS mutated
MeSH Terms: conditions — Colorectal Neoplasms | interventions — folfirinox; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Folfirinox-R (Experimental): Folfirinox + regorafenib
  Interventions: Combination Product: Folfirinox + regorafenib

INTERVENTIONS:
Combination Product: Folfirinox + regorafenib — folfirinox : from day 1 to day 3 regorafenib : day 4 to day 10 a cycle during 14 days

SUMMARY:
Safety, tolerability and efficacy of regorafenib in combination with FOLFIRINOX in patients with RAS-mutated metastatic colorectal cancer: a dose-escalation, phase I/II trial

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a major cause of morbidity and mortality globally. More than 50% of patients can be expected to develop metastatic disease, and most of these patients will require palliative systemic therapy. The primary goal for patients who present with technically resectable liver metastases is definitely cure, with R0 resection as the primary goal. Consequently, any patient with limited liver and/or lung metastases should be considered a candidate for potential secondary resection as there are no criteria that allow physicians to distinguish between those patients for whom purely palliative treatment and those or whom potentially curative treatment is appropriate. Although survival times are slightly shorter for patients who undergo conversion therapy followed by surgery than for patients with initially resectable metastatic disease, they are far better than if resection is not carried out at all. First-line therapy commonly involves the doublet regimens of 5-fluorouracil, folinic acid, and either oxaliplatin or irinotecan. The addition of targeted therapies, such as bevacizumab (a pure anti-angiogenic agent which binds circulating VEGF-A), cetuximab, and panitumumab, to FOLFOX (5FU, oxaliplatin) or FOLFIRI (5FU, irinotecan) may be helpful to some patients in improving tumor response and ultimately overall survival. The cytotoxic triplet FOLFOXIRI (5FU, oxaliplatin, irinotecan) with or without bevacizumab may be an option in selected fit and motivated patients when cytoreduction (tumour shrinkage) is needed to undergo conversion therapy.

RAS mutations are found in about 50% of mCRC tumors. These mutations exclude affected patients from epidermal growth factor receptor (EGFR)-directed therapy. Besides their negative predictive value, RAS mutations may also carry distinct prognostic information. Modest studied the prognosis by RAS status of a total of 1239 mCRC patients from five randomized trials studying 2-CT. Actually, PFS and OS were significantly influenced by molecular subgroups. Multivariate comparison of Progression-Free Survival (PFS) and Overall Survival (OS) in patients with mutant tumors versus patients with non-mutated tumors revealed a negative prognostic effect of RAS mutations. Interestingly, the negative prognostic role of these mutations was consistently observed across different treatment regimens (subgroups of irinotecan- and oxaliplatin-treated patients as well as in bevacizumab- and non-bevacizumab-treated patients). Median PFS and OS were 10.3 vs. 9.5 months and 26.9 vs. 21.1 months in RAS-wildtype (and BRAF-wildtype) and RAS-mut patients, respectively. The TRIBE consortium reported that a 3-CT (FOLFOXIRI) combined with bevacizumab provided a significantly longer PFS (the primary end-point of the study) than did the 2-CT FOLFIRI plus bevacizumab . In the subgroup of RAS- and BRAF-wild-type patients, those in the FOLFOXIRI plus bevacizumab group reported a median PFS of 13.7 months (95% CI, 10.1-18.1) compared with 12.2 months (95%CI, 9.5-14.4) in the FOLFIRI plus bevacizumab group (HR 0.85, 95%CI 0.55-1.3).

Later on, the same group reported that FOLFOXIRI plus bevacizumab provided a significantly longer overall survival than the FOLFIRI plus bevacizumab group (HR 0.80, 95%CI 0·65-0·98; p=0·03) . Looking at survival by RAS status, Cremolini reported that median OS was 37.1 months (95%CI, 29.7-42.7) in the RAS- and BRAF-wild-type subgroup compared with 25.6 months (95%CI, 22.4-28.6) in the RAS-mut subgroup (HR 1.49, 95%CI, 1.11-1·99). Interestingly, median PFS was 13.7 months (95% CI 10.1-18.1) in the RAS-wild-type subgroup treated with FOLFOXIRI plus bevacizumab, while PFS data were not given for the RAS-mut patients . However, for these RAS-mut patients, it was possible to estimate the median PFS (i.e. 9.4 months) from the Kaplan-Meier curve which was provided.

Regorafenib is a small-molecule inhibitor of multiple membrane-bound and intracellular kinases. Beyond its well-known antiangiogenic properties, regorafenib has also less-known anti-proliferative activities in human colon cancer cell lines. Interestingly, regorafenib potently inhibits growth of patient-derived CRC xenografts alone and in combination with irinotecan . Regorafenib is approved for refractory mCRC patients, for locally advanced, unresectable or metastatic GIST patients and for HCC patients previously treated with sorafenib. The recommended dose is 160 mg (40 mg × 4 tablets) orally, once daily for the first 21 days of each 28-day cycle. Two phase III trials demonstrated a significant overall survival benefit for regorafenib over placebo in patients with mCRC who progressed on standard therapies . Two phase II trials studied the safety and efficacy profile of regorafenib when combined to chemotherapy in patients with mCRC . In vitro data indicate that both regorafenib and its metabolite M-2 inhibit glucuronidation mediated by UGT1A1 ( uridine 5'diphospho-glucuronosyl transferase A1) and UGT1A9 (whereas M-5 only inhibits UGT1A1), hence triggering potential pharmacokinetic interactions. The study from Schultheis was designed to explore whether addition of regorafenib to FOLFOX or FOLFIRI could be feasible as a treatment of mCRC, in terms of safety and pharmacokinetic interactions of the various drug components of the regimen. Forty-five patients were treated every 2 weeks with 5-fluorouracil 400 mg/m² bolus then 2400 mg/m² over 46 h, folinic acid 400 mg/m², and either oxaliplatin 85 mg/m² or irinotecan 180 mg/m².

On days 4-10, patients received regorafenib 160 mg orally once daily. Drug-related adverse events resulted in dose modification, dose interruption, or permanent discontinuation of study treatment in 31 (69%) patients overall (18 [72%] FOLFOX and 13 [65%] FOLFIRI).

Dose reduction or dose interruption of at least one of the chemotherapy components was observed in 52% of patients treated with FOLFOX and 65% of patients receiving FOLFIRI. A dose reduction of 5-fluorouracil due to AEs was necessary in 18% of administered cycles. 5-Fluorouracil administration was omitted in 8% of cycles. Oxaliplatin and irinotecan doses were reduced in 11% and 12% and interrupted in 11% and 5% of administered cycles, respectively. Actually, regorafenib had acceptable tolerability in combination with chemotherapy. The most frequent grade 3-4 AEs were: neutropenia (45%), Hand-Foot Skin Reaction (15%), diarrhea (10%), and hypophosphatemia (12%). Regarding pharmacokinetics, area under the curve (AUC) of irinotecan was significantly higher in cycle 2 (following regorafenib dosing) than in cycle 1 (before regorafenib dosing); the ratio of AUC values (cycle 2:cycle 1) was 1.28 (90% confidence interval [CI] 1.06 -1.54). Cmax of irinotecan was only slightly increased, and t½ (half-life) was unchanged. For SN-38 (metabolite of irinotecan), AUC was significantly higher in cycle 2 than in cycle 1 (ratio 1.44, 90% CI 1.12-1.85), while Cmax was unchanged. In line with the known elimination pathways of platinum and 5-fluorouracil, no pharmacokinetic interaction with regorafenib was seen . The study from O'Neil was designed to show whether the addition of regorafenib to FOLFIRI improves PFS (over a placebo-FOLFIRI arm) when given as second-line therapy for patients treated initially with oxaliplatin and fluoropyrimidine-based therapy. The regorafenib/FOLFIRI schedule that was used was the one proposed by Schultheis (i.e. standard FOLFIRI with irinotecan 180 mg/m² plus regorafenib 160 mg daily from day 4 to 10). The study met its primary endpoint of demonstrating that the addition of regorafenib to FOLFIRI prolongs PFS compared to FOLFIRI alone with a HR (Hazard Ratio) of 0.72. When looking at tumor response, authors found that regorafenib (combined to chemo) provided more partial responses than placebo plus chemo (35% vs. 19%, p= 0.045). The combination was very tolerable, with little increase in toxicity compared to the control chemotherapy regimen. Of note, regarding the top-3 reported severe (gr. 3-4) AEs, neutropenia, diarrhea, and hypophosphatemia were reported in 41%, 15%, and 14% of the patients, respectively (as compared to 30%, 5%, and 0% in the placebo group).

Actually, there is room to combine regorafenib with a chemo triplet such as FOLFIRINOX (5-fluorouracil, irinotecan, oxaliplatin) on the following conditions: controlling patients on UGT1A polymorphisms (at least UGT1A1), stepwise dose-escalation of irinotecan and regorafenib, mandatory granulocyte growth-factor injections.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for full study.
2. Documentation of tumor RAS mutation, wild-type homozygous, heterozygous status of UGT1A1 gene. The status of UGT1A1 gene will be performed by the laboratory chosen by the investigator
3. Serum uracile < 16 ng/ml
4. Measurable disease, defined as at least one unidimensional measurable lesion on a CT scan, according to RECIST version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
6. Life expectancy of at least 3 months.
7. Adequate bone marrow, renal and liver functions as evidenced by the following laboratory requirements within 7 days prior to study treatment initiation: Absolute neutrophil count (ANC) ≥ 1,500/ mm3 without biologic response modifiers such as granulocyte colony-stimulating factor (G-CSF), within 21 days before the start of study treatment, Platelet count ≥ 100 000/mm3 , without platelet transfusion within 21 days before the start of study treatment ,Hemoglobin (Hb) ≥ 9 g/dL, without blood transfusion or erythropoietin, within 21 days before the start of study treatment, Serum creatinine ≤ 1.5 x upper limit of normal(ULN) Serum calcium ≥ Lower limits of normal LLN and ≤ 1.2 x UNL ; Serum magnesium ≥ LLN and ≤ 1.2 x UNL ; Kalemia ≥ LLN, Glomerular filtration rate as assessed by the estimated glomerular filtration rate (eGFR) ≥ 50 mL/min per 1.73 m2 calculated by the Modification of Diet in Renal Disease (MDRD) abbreviated formula, Total bilirubin ≤ 1.5 x ULN, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer), Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5.0 x ULN for patients with liver involvement for their cancer and/or bone metastases).
8. Lipase ≤ 1.5 x ULN.
9. Adequate coagulation, as assessed by the following laboratory test results:

   International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 x ULN, Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN, Note: Patients on stable dose (dose has not been changed in at least 28 days) of anticoagulation therapy will be allowed to participate if they have no sign of bleeding or clotting and INR / PT and PTT / aPTT test results are compatible with the acceptable benefit-risk ratio at the investigator's discretion. In such case, limits as noted would not apply.
10. For women of reproductive potential, negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test obtained within 7 days before the start of study treatment. Women not of reproductive potential are female patients who are postmenopausal or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy).
11. For women of childbearing potential and men, agreement to use an adequate contraception for the duration of study participation and up to 4 months following completion of therapy for women and 6 months for male patients. Females of childbearing potential who are sexually active with a non-sterilized male partner must use 2 methods of effective contraception. The investigator or a designated associate is requested to advise the patient on how to achieve an adequate birth control.

    Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.
12. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
13. Affiliation to the Social Security System.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to study inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (noninvasive tumor), Tis (carcinoma in situ) and T1 (lamina propria invasion)].
2. Discovery of metastases within 6 months after the termination of adjuvant chemotherapy.
3. Previous treatment for metastatic disease. Radiotherapy within 28 days prior to first dose of treatment.
4. Active cardiac disease including any of the following:

   Congestive heart failure New York Heart Association (NYHA) class 2, Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), Myocardial infarction less than 6 months before first dose of treatment, Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
5. ECG with a QT/QTc interval higher than 450 ms for men and higher than 470 ms for women Uncontrolled hypertension.
6. Uncontrolled hypertension. (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
7. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before start of treatment.

8;Persistent proteinuria of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE V5) grade 3 (i.e. urinary protein ≥ 3.5 g/24 hrs) 9;Peripheral neuropathy > grade1 (NCI-CTCAE v5). 10.Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to first dose of Treatment.

11.Ongoing infection >grade 2 (NCI-CTCAE v5). 12.Known history of human immunodeficiency virus (HIV) infection. 13.Chronic hepatitis B or C infection (if hepatitis status cannot be obtained from medical records, re-testing is required).

14.Seizure disorder requiring medication. 15.Symptomatic metastatic brain or meningeal tumors. 16.Evidence or history of any bleeding diathesis, irrespective of severity. Any hemorrhage or bleeding event ≥ grade 3 (NCI-CTCAE v5) within 4 weeks prior to the start of study medication.

17.History of organ allograft. 18.Non-healing wound, ulcer, or bone fracture. 19.Dehydration Grade 1 NCI-CTCAE v5). 20.Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.

21.Known hypersensitivity to any of the study drugs, study drug classes, or any constituent of the products.

22.Interstitial lung disease with ongoing signs and symptoms. 23.Concomitant intake of St. John's wort. 24.Live attenuated vaccines are prohibited 10 days before the treatment, during the treatment and 3 months after the termination of treatment 25.History of gastrointestinal fistula or perforation 26.Inability to swallow oral medication. 27.Any malabsorption condition. 28.Pregnant or breast-feeding subjects. 29.Any condition that, in the opinion of the investigator, would interfere with the evaluation of study treatment or interpretation of patient safety or study results.

30.Participation in another clinical study with an investigational product during the last 30 days before inclusion. 31.Patients who might be interconnected with or dependent on the sponsor site or the investigator.

32.Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Adenis, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (4):
- France (4):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - Centre Georges-François Leclerc, Dijon, Côte d'Or
  - Centre Cario - HPCA, Plérin, Finistère
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan, the clinical study report and the analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Access to study data upon written detailed request sent to Institute of Montpellier Cancer after publication.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from Institute of Montpellier Cancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Modest DP, Ricard I, Heinemann V, Hegewisch-Becker S, Schmiegel W, Porschen R, Stintzing S, Graeven U, Arnold D, von Weikersthal LF, Giessen-Jung C, Stahler A, Schmoll HJ, Jung A, Kirchner T, Tannapfel A, Reinacher-Schick A. Outcome according to KRAS-, NRAS- and BRAF-mutation as well as KRAS mutation variants: pooled analysis of five randomized trials in metastatic colorectal cancer by the AIO colorectal cancer study group. Ann Oncol. 2016 Sep;27(9):1746-53. doi: 10.1093/annonc/mdw261. Epub 2016 Jun 29. PMID 27358379
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- [Background] Schmieder R, Hoffmann J, Becker M, Bhargava A, Muller T, Kahmann N, Ellinghaus P, Adams R, Rosenthal A, Thierauch KH, Scholz A, Wilhelm SM, Zopf D. Regorafenib (BAY 73-4506): antitumor and antimetastatic activities in preclinical models of colorectal cancer. Int J Cancer. 2014 Sep 15;135(6):1487-96. doi: 10.1002/ijc.28669. Epub 2014 Apr 17. PMID 24347491
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Background] Schultheis B, Folprecht G, Kuhlmann J, Ehrenberg R, Hacker UT, Kohne CH, Kornacker M, Boix O, Lettieri J, Krauss J, Fischer R, Hamann S, Strumberg D, Mross KB. Regorafenib in combination with FOLFOX or FOLFIRI as first- or second-line treatment of colorectal cancer: results of a multicenter, phase Ib study. Ann Oncol. 2013 Jun;24(6):1560-7. doi: 10.1093/annonc/mdt056. Epub 2013 Mar 13. PMID 23493136
- [Background] Leitinger B. Discoidin domain receptor functions in physiological and pathological conditions. Int Rev Cell Mol Biol. 2014;310:39-87. doi: 10.1016/B978-0-12-800180-6.00002-5. PMID 24725424
- [Background] Rammal H, Saby C, Magnien K, Van-Gulick L, Garnotel R, Buache E, El Btaouri H, Jeannesson P, Morjani H. Corrigendum: Discoidin Domain Receptors: Potential Actors and Targets in Cancer. Front Pharmacol. 2016 Sep 30;7:346. doi: 10.3389/fphar.2016.00346. eCollection 2016. PMID 27703433
- [Background] Gao H, Chakraborty G, Zhang Z, Akalay I, Gadiya M, Gao Y, Sinha S, Hu J, Jiang C, Akram M, Brogi E, Leitinger B, Giancotti FG. Multi-organ Site Metastatic Reactivation Mediated by Non-canonical Discoidin Domain Receptor 1 Signaling. Cell. 2016 Jun 30;166(1):47-62. doi: 10.1016/j.cell.2016.06.009. PMID 27368100
- [Background] Jeitany M, Leroy C, Tosti P, Lafitte M, Le Guet J, Simon V, Bonenfant D, Robert B, Grillet F, Mollevi C, El Messaoudi S, Otandault A, Canterel-Thouennon L, Busson M, Thierry AR, Martineau P, Pannequin J, Roche S, Sirvent A. Inhibition of DDR1-BCR signalling by nilotinib as a new therapeutic strategy for metastatic colorectal cancer. EMBO Mol Med. 2018 Apr;10(4):e7918. doi: 10.15252/emmm.201707918. PMID 29438985
- [Background] Zopf D, Fichtner I, Bhargava A, Steinke W, Thierauch KH, Diefenbach K, Wilhelm S, Hafner FT, Gerisch M. Pharmacologic activity and pharmacokinetics of metabolites of regorafenib in preclinical models. Cancer Med. 2016 Nov;5(11):3176-3185. doi: 10.1002/cam4.883. Epub 2016 Oct 13. PMID 27734608
- [Background] Mouliere F, El Messaoudi S, Gongora C, Guedj AS, Robert B, Del Rio M, Molina F, Lamy PJ, Lopez-Crapez E, Mathonnet M, Ychou M, Pezet D, Thierry AR. Circulating Cell-Free DNA from Colorectal Cancer Patients May Reveal High KRAS or BRAF Mutation Load. Transl Oncol. 2013 Jun 1;6(3):319-28. doi: 10.1593/tlo.12445. Print 2013 Jun. PMID 23730412
- [Background] Mouliere F, El Messaoudi S, Pang D, Dritschilo A, Thierry AR. Multi-marker analysis of circulating cell-free DNA toward personalized medicine for colorectal cancer. Mol Oncol. 2014 Jul;8(5):927-41. doi: 10.1016/j.molonc.2014.02.005. Epub 2014 Mar 24. PMID 24698732
- [Background] Thierry AR, Mouliere F, El Messaoudi S, Mollevi C, Lopez-Crapez E, Rolet F, Gillet B, Gongora C, Dechelotte P, Robert B, Del Rio M, Lamy PJ, Bibeau F, Nouaille M, Loriot V, Jarrousse AS, Molina F, Mathonnet M, Pezet D, Ychou M. Clinical validation of the detection of KRAS and BRAF mutations from circulating tumor DNA. Nat Med. 2014 Apr;20(4):430-5. doi: 10.1038/nm.3511. Epub 2014 Mar 23. PMID 24658074
- [Background] Thierry AR, El Messaoudi S, Mollevi C, Raoul JL, Guimbaud R, Pezet D, Artru P, Assenat E, Borg C, Mathonnet M, De La Fouchardiere C, Bouche O, Gavoille C, Fiess C, Auzemery B, Meddeb R, Lopez-Crapez E, Sanchez C, Pastor B, Ychou M. Clinical utility of circulating DNA analysis for rapid detection of actionable mutations to select metastatic colorectal patients for anti-EGFR treatment. Ann Oncol. 2017 Sep 1;28(9):2149-2159. doi: 10.1093/annonc/mdx330. PMID 28911069
- [Background] Tie J, Kinde I, Wang Y, Wong HL, Roebert J, Christie M, Tacey M, Wong R, Singh M, Karapetis CS, Desai J, Tran B, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA as an early marker of therapeutic response in patients with metastatic colorectal cancer. Ann Oncol. 2015 Aug;26(8):1715-22. doi: 10.1093/annonc/mdv177. Epub 2015 Apr 7. PMID 25851626
- [Background] Vidal J, Muinelo L, Dalmases A, Jones F, Edelstein D, Iglesias M, Orrillo M, Abalo A, Rodriguez C, Brozos E, Vidal Y, Candamio S, Vazquez F, Ruiz J, Guix M, Visa L, Sikri V, Albanell J, Bellosillo B, Lopez R, Montagut C. Plasma ctDNA RAS mutation analysis for the diagnosis and treatment monitoring of metastatic colorectal cancer patients. Ann Oncol. 2017 Jun 1;28(6):1325-1332. doi: 10.1093/annonc/mdx125. PMID 28419195
- [Background] Thierry AR, Pastor B, Jiang ZQ, Katsiampoura AD, Parseghian C, Loree JM, Overman MJ, Sanchez C, Messaoudi SE, Ychou M, Kopetz S. Circulating DNA Demonstrates Convergent Evolution and Common Resistance Mechanisms during Treatment of Colorectal Cancer. Clin Cancer Res. 2017 Aug 15;23(16):4578-4591. doi: 10.1158/1078-0432.CCR-17-0232. Epub 2017 Apr 11. PMID 28400427
- [Derived] Adenis A, Ghiringhelli F, Gauthier L, Mazard T, Evesque L, Evrard A, Chalbos P, Moussion A, Gourgou S, Ychou M. Regorafenib plus FOLFIRINOX as first-line treatment for patients with RAS-mutant metastatic colorectal cancer (FOLFIRINOX-R trial): a dose-escalation study. Cancer Chemother Pharmacol. 2024 Sep;94(3):443-452. doi: 10.1007/s00280-024-04682-4. Epub 2024 Jul 10. PMID 38987363
- [Derived] Adenis A, Mazard T, Fraisse J, Chalbos P, Pastor B, Evesque L, Ghiringhelli F, Mollevi C, Delaine S, Ychou M. FOLFIRINOX-R study design: a phase I/II trial of FOLFIRINOX plus regorafenib as first line therapy in patients with unresectable RAS-mutated metastatic colorectal cancer. BMC Cancer. 2021 May 17;21(1):564. doi: 10.1186/s12885-021-08312-7. PMID 34001059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from 14/05/2019 to 15/10/2021.
Pre-assignment Details: Screening based on Uridine diphosphate-GlucuronosylTransferase (UGT1A1) status and DiHydroPyrimidine Dehydrogenase (DHPD) status with serum uracile < 16 ng/ml.
Groups:
- Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg (PO): Cohort 1: Participants were administered 150 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products is unchanged. Oxaliplatin, 5 FU Bolus and 5FU continuous are at 85 mg/m², 400 mg/m² and 2400 mg/m² respectively.
- Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg (PO): Cohort 2: Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib.
  The dosage of the others products is unchanged. Oxaliplatin, 5FU Bolus and 5FU continuous are at 85 mg/m², 400 mg/m² and 2400 mg/m² respectively.
- Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg (PO): Cohort 3: Participants were administered 180 mg/m² of Irinotecan and 160 mg of Regorafenib.
  The dosage of the others products is unchanged. Oxaliplatin, 5 FU Bolus and 5FU continuous are at 85 mg/m², 400 mg/m² and 2400 mg/m² respectively.
Period: Overall Study
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg (PO)
Started | 3 | 6 | 4
Completed | 3 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg/m² (PO): Cohort 1 : Participants were administered 150 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged i.e Oxaliplation at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg/m² (PO): Cohort 2: Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged i.e Oxaliplation at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg/m² (PO): Cohort 3: Participants were administered 180 mg/m² of Irinotecan and 160 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged i.e Oxaliplation at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Total: Total of all reporting groups
Arm/Group | Experimental Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg/m² (PO) | Experimental Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg/m² (PO) | Experimental Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg/m² (PO) | Total
Number analyzed (Participants) | 3 | 6 | 4 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [49 to 65] | 69 [40 to 76] | 64.5 [49 to 76] | 65 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 1 | 3 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 6 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 3 | 6 | 4 | 13
Assessment of the patient's general condition using the ECOG scale [Number; unit: participants] — The physician determines the general condition of patient by using the scale ECOG.
  ECOG 0 : Fully active patient, able to perform the same pre-morbid activities without restriction. Very good general condition.
  ECOG 1 : Patient restricted in physical activities, but ambulatory and able to perform light or sedentary activities, e.g. light housework or administrative tasks. Good general condition.
  participants
    0 | 1 | 2 | 3 | 6
    1 | 2 | 4 | 1 | 7
Weight [Median (Inter-Quartile Range); unit: Kilograms] | 71 [65 to 95] | 69 [42 to 96] | 78 [57 to 106] | 69 [42 to 106]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m²] | 22.9 [21.5 to 29] | 27.2 [16 to 34] | 24.3 [19.7 to 31.7] | 27 [16 to 34]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mm/hg] | 130 [120 to 140] | 127 [113 to 146] | 140.5 [133 to 158] | 130 [113 to 158]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mm/hg] | 84 [67 to 89] | 73 [64 to 87] | 82 [73 to 85] | 79 [64 to 89]
Tumor location [Number; unit: participants]
  Right colon | 1 | 1 | 0 | 2
  Left colon | 0 | 1 | 0 | 1
  Transverse colon | 0 | 1 | 0 | 1
  Recto-sigmoid junction | 0 | 1 | 1 | 2
  Rectum | 2 | 2 | 3 | 7
Lymph node dissection [Count of Participants; unit: Participants]
  Lymph node dissection done | 3 | 5 | 3 | 11
  Lymph node dissection not done | 0 | 1 | 1 | 2
Adenocarcinoma type [Count of Participants; unit: Participants]
  well/moderately differentiated | 1 | 4 | 0 | 5
  Poorly differentiated/undifferentiated | 0 | 2 | 4 | 6
  Unknown | 2 | 0 | 0 | 2
Depth of tumoral invasion in the wall of colon/rectum determined by pathologist [Count of Participants; unit: Participants] — T1: The cancer has grown through the muscularis mucosa into the submucosa. Locally advanced tumor. Very good pronostic.
  T2 : The cancer have grown into the muscularis propria. Good pronostic. T3: The cancer has grown into the outermost layers of the colon or rectum but has not gone through them. Bad pronostic.
  T4a: The cancer has grown through the wall of the colon or rectum but has not grown into other organs. Very bad pronostic.
  T4b: The cancer has grown through the wall of the colon or rectum and is attached to or has grown into other nearby tissues or organs.Very bad pronostic.
  Participants
    T3 | 0 | 1 | 1 | 2
    T4b | 0 | 1 | 0 | 1
    TX (not operated) | 2 | 4 | 3 | 9
    Unknown | 1 | 0 | 0 | 1
Comparison of number of patients with positive nodes versus negative nodes [Count of Participants; unit: Participants] — N0 means there are no lymph nodes containing cancer cells.Very good prognosis. N1 means there are cancer cells in 1 to 3 lymph nodes. Intermediate prognosis. N2 means means there are cancer cells in more than 4 lymph nodes.Bad prognosis.
  Participants
    N0 | 0 | 0 | 1 | 1
    N1 | 0 | 2 | 1 | 3
    N2 | 0 | 1 | 0 | 1
    NX (not operated) | 2 | 3 | 2 | 7
    Unknown | 1 | 0 | 0 | 1
Comparison of number of metastatic patients versus metastasis-free patients [Count of Participants; unit: Participants] — M0 : metastasis-free patient. Good prognosis. M1: metastatic patient. Bad prognosis.
  Participants
    M0 | 0 | 1 | 1 | 2
    M1 | 3 | 5 | 2 | 10
    M1a | 0 | 0 | 1 | 1
Metastatic location [Number; unit: metastatic sites]
  Brain | 0 | 1 | 0 | 1
  Liver | 3 | 5 | 4 | 12
  Lymphatic nodes | 0 | 2 | 1 | 3
  Bone | 0 | 0 | 0 | 0
  Lung | 1 | 3 | 1 | 5
  Peritoneum | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pre-specified Treatment-related Adverse Events
Description: The physician determines pre-specified treatment-related toxicities and grades them by using the Common Terminology Criteria for Adverse Events (NCI-CTC Version 5). 1 - Mild: 2 - Moderate: 3 - Severe: 4 - Life-threatening: 5 - Death.
  Th evaluation is realized during the first three cycles.
Time Frame: At the end of cycle 1 to 3 (each cycle is 14 days)
Population: Evaluable population for Dose-limiting toxicity (DLT). The list of DLTs is pre-specified in the protocol.
Measure: Number; unit: participants
Groups:
- Experimental: Irinotecan 150 mg/m² and Regorafenib 120 mg: Cohort 1: Participants were administered 150 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental : Irinotecan 180 mg/m² and Regorafenib 120 mg: Cohort 2 : Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental : Irinotecan 180 mg/m² and Regorafenib 160 mg: Cohort 3 : Participants were administered 180 mg/m² of Irinotecan and 160 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
Arm/Group | Experimental: Irinotecan 150 mg/m² and Regorafenib 120 mg | Experimental : Irinotecan 180 mg/m² and Regorafenib 120 mg | Experimental : Irinotecan 180 mg/m² and Regorafenib 160 mg
Number analyzed (Participants) | 3 | 6 | 4
participants | 3 | 5 | 3

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from date of inclusion to date of first observed disease progression (investigator's radiological or clinical assessment) or death due to any cause, if death occurs before progression is documented. . A central review of CT-scans is planned for patients found progression-free at 48 weeks. Patients without tumor progression or death at the time of analysis will be censored at their last date of tumor assessment.
Time Frame: From baseline of patient until the first observed disease progression
Population: Intention to treat
Measure: Median (Full Range); unit: Month
Groups:
- Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO): Cohort 1: Participants were administered 150 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatin at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO): Cohort 2: Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatin at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO): Cohort 3: Participants were administered 180 mg/m² of Irinotecan and 160 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatin at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 3 | 6 | 4
Month | 12.5 [8.7 to 15.4] | 8.2 [3.1 to 9.1] | 5.1 [3.4 to 7.7]

3. Secondary Outcome: Number of Patients With Disease Control
Description: The disease control corresponds to stable, partial and complete responses determined by RECIST criteria.
  Criteria recist are based on lesions measurement determined by radiologist. Calculation : the values at the baseline minus the lowest values (nadir)
Time Frame: Up to 6 months, from baseline of patient to the point where the values are the lowest (nadir).
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 3 | 6 | 4
Participants | 3 | 6 | 4

4. Secondary Outcome: Number of Participants With Objective Response
Description: The objective response corresponds to partial and complete responses determined by RECIST criteria.
  Criteria recist are based on lesions measurement determined by radiologist. Calculation : The values at the baseline minus the lowest values (nadir)
Time Frame: Up to 6 months, from baseline of patient to the point where the values are the lowest (nadir).
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 3 | 6 | 4
participants | 2 | 3 | 4

5. Secondary Outcome: Overall Survival (OS)
Time Frame: From baseline to date of patient death
Population: Intention to treat
Measure: Median (Full Range); unit: Month
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 3 | 6 | 4
Month | 16.7 [15.6 to 18] | 13.3 [7 to 20] | 10.7 [7.2 to 15]

6. Secondary Outcome: The Median of Regression of Tumor Size
Description: The percentage of regression of tumor size to its lowest value (nadir), compared with the pre-treatment tumor size (baseline), according to RECIST criteria (this is the reference method for evaluating cancer treatments based on the measurement of lesions by radiologist).
Time Frame: Up to 6 months, from baseline of patient to the point where the values are the lowest (nadir).
Population: Intention to treat
Measure: Median (Full Range); unit: Percentage
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 3 | 6 | 4
Percentage | 55.3 [21.7 to 64.7] | 40.85 [1.1 to 61.7] | 60.75 [40.6 to 73]

7. Secondary Outcome: Maintenance Treatment With Regorafenib Alone
Description: Description by cycles of Regorafenib maintenance treatment after 12 cycles of Folfirinox-R
Time Frame: Up to 16 weeks (after 12 cycles of Folfirinox-R)
Population: Population by step and evaluable for safety
Measure: Count of Participants; unit: Participants
Arm/Group | Folfirinox-R
Number analyzed (Participants) | 13
Participants
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: number analyzed (Participants) | 3
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: 2 cycles received | 0
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: 3 cycles received | 0
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: 4 cycles received | 0
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: 6 cycles received | 0
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: 8 cycles received | 0
  Step 1 : IRINOTECAN 150 / REGORAFENIB 120: No cycles received | 3
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: number analyzed (Participants) | 6
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: 2 cycles received | 1
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: 3 cycles received | 0
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: 4 cycles received | 1
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: 6 cycles received | 0
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: 8 cycles received | 1
  Step 2 : IRINOTECAN 180 / REGORAFENIB 120: No cycles received | 3
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: number analyzed (Participants) | 4
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: 2 cycles received | 0
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: 3 cycles received | 1
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: 4 cycles received | 0
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: 6 cycles received | 1
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: 8 cycles received | 0
  Step 3 : IRINOTECAN 180 / REGORAFENIB 160: No cycles received | 2
  All steps: 2 cycles received | 1
  All steps: 3 cycles received | 1
  All steps: 4 cycles received | 1
  All steps: 6 cycles received | 1
  All steps: 8 cycles received | 1
  All steps: No cycles received | 8

8. Secondary Outcome: Determination of Circulating Free DNA Concentration (Not Available)
Description: From baseline of first patient until the end of treatment
Time Frame: Baseline, 8 weeks, 16 weeks etc. through the end of treatment
Population: Blood samples were not analyzed because the number of patients per cohort was too low. Consequently, the data is not available and cannot be populated.
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Resection (R) Rates (Not Available)
Description: Through the treatment
Time Frame: Approximately at 6 months
Population: as for outcome 8
Groups:
- Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg (PO): Cohort 1: Participants were administered 150 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental : Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg (PO): Cohort 2 : Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
- Experimental : Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg (PO): Cohort 3 : Participants were administered 180 mg/m² of Irinotecan and 160 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatine at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib 120 mg (PO) | Experimental : Irinotecan 180 mg/m² (IV) and Regorafenib 120 mg (PO) | Experimental : Irinotecan 180 mg/m² (IV) and Regorafenib 160 mg (PO)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the baseline up to one month after the last cycle of chemotherapy, up to 7 months (AE ans SAEs). From the baseline up to 20 months for all-cause mortality.
Groups:
- Experimental: Irinotecan 180 mg/m² (IV) Cand Regorafenib at 120 mg (PO): Cohort 2: Participants were administered 180 mg/m² of Irinotecan and 120 mg of Regorafenib every 14 days.
  The dosage of the others products are unchanged. Oxaliplatin at 85 mg/m², 5FU Bolus at 400 mg/m² and 5FU continuous at 2400 mg/m².
Arm/Group | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) Cand Regorafenib at 120 mg (PO) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO)
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/6 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) (N=3) | Experimental: Irinotecan 180 mg/m² (IV) Cand Regorafenib at 120 mg (PO) (N=6) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO) (N=4)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal subocclusive syndrom (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Irinotecan 150 mg/m² (IV) and Regorafenib at 120 mg (PO) (N=3) | Experimental: Irinotecan 180 mg/m² (IV) Cand Regorafenib at 120 mg (PO) (N=6) | Experimental: Irinotecan 180 mg/m² (IV) and Regorafenib at 160 mg (PO) (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (8) | 2 (4)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aphtous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (8) | 6 (25) | 4 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (11) | 4 (7)
Rectal syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (1) | 2 (4)
Asthenia (General disorders) | 2 (9) | 6 (12) | 3 (10)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Erythema induratum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis E (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood alcaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactatce dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Gammaglutamyl transferase increased (Investigations) | 0 (0) | 1 (1) | 2 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (4) | 3 (4) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (13) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Distal wekness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgueusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (3) | 4 (7) | 3 (9)
Palmar-plantar erythrodysaesthesia syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 4 (6) | 4 (24)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Transaminase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03828799/Prot_SAP_000.pdf